CLINICAL TRIAL: NCT01773811
Title: Effects of Narrative Writing Duration and Post-writing Processing Instructions on PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMO-0004
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder (PTSD); Narrative Writing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Individuals will write objectively about the events of their day.
- Narrative Writing: Trauma-Assigned (Experimental): Trauma-assigned: Individuals will write about their most traumatic life experience and be instructed to continue to think about their writing topic in the weeks following writing.
  Interventions: Behavioral: Narrative Writing: Trauma-Assigned
- Narrative Writing: Trauma-Spontaneous (Active Comparator): Individuals will write about their most traumatic life experience but will not be given further instructions for processing. Any additional processing about their writing topic in the weeks following writing will be considered spontaneous.
  Interventions: Behavioral: Narrative Writing: Trauma-Spontaneous

INTERVENTIONS:
Behavioral: Narrative Writing: Trauma-Assigned — Individuals will be writing about their most traumatic life event for 3 consecutive days for 20 minutes each. Those in the assigned group will be given instructions and weekly reminders to continue to think about their most traumatic event.
  Arms: Narrative Writing: Trauma-Assigned
Behavioral: Narrative Writing: Trauma-Spontaneous — Individuals will be writing about their most traumatic life event for 3 consecutive days for 20 minutes each. Those in the spontaneous group will be given no further instructions.
  Arms: Narrative Writing: Trauma-Spontaneous

SUMMARY:
The current study proposes to directly measure how processing after participating in written disclosure about a traumatic life event affects physical and psychological outcomes.

DETAILED DESCRIPTION:
Previous research has established the potential for narrative writing about traumatic events to result in positive benefits for physical and psychological health. Research has also provided evidence that written disclosure may reduce post-traumatic stress disorder (PTSD) symptoms. Several mechanisms of action have been proposed to explain why written disclosure produces positive benefits, but all have focused on processes occurring during the writing session. It has been suggested, however, that additional processing may occur after the writing exercises are over, yet no research has studied the influence of this processing on outcomes. The current study proposes to directly measure how processing after participating in written disclosure affects physical and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a traumatic life event (DSM-IV-TR Criterion A)
* Currently experiencing clinically significant levels of PTSD symptoms

Exclusion Criteria:

* Currently receiving psychotherapy
* On medication that is not stable (i.e. medication has been changed within the past 6 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Level of PTSD symptoms as measured by the Clinician Administered PTSD Scale | 1 month after final writing session

SECONDARY OUTCOMES:
Physical health | 1 month after final writing session
  Physical health as measured by the Pennebaker Inventory of Limibic Languidness (PILL)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lombardo, PhD, Principal Investigator — University of Mississippi, Oxford
Locations (1):
- The University of Mississippi, University, Mississippi, United States